CLINICAL TRIAL: NCT04967651
Title: Analysis of Risk Factors and Establishment and Application of a Clinical Early Warning Model for Postoperative Pulmonary Complications in Patients Undergoing Cardiac Surgery
Brief Title: Analysis of Risk Factors and Establishment of Early Warning Model for Pulmonary Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Central Hospital (Other); Shanxi Cardiovascular Hospital (Other); Qinghai People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PPC202106
Record Dates: First submitted 2021-07-15; First posted 2021-07-19 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pulmonary Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pulmonary complications following cardiac surgery
- Patients without pulmonary complications following cardiac surgery

SUMMARY:
The purpose of this study is to collect perioperative diagnosis and treatment information for cardiac surgery patients, collect blood samples for laboratory testing when necessary, and analyze the data to clarify the risk factors of pulmonary complications in patients undergoing cardiac surgery during the perioperative period. On this basis, a clinical early warning model for pulmonary complications after cardiac surgery will be developed to reduce the risk of pulmonary complications and even death in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older;
* Elective cardiac surgery under general anesthesia

Exclusion Criteria:

* Patients and their family members refused to be enrolled;
* Patients unable to communicate due to language barriers such as dementia;
* Patients admitted to ICU 24h before surgery;
* Estimated duration of surgery less than 2 hours;
* Patients died or discharged within 24 hours after surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who planned elective cardiac surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The occurrence of postoperative pulmonary complications | 1 week after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, China